CLINICAL TRIAL: NCT06872125
Title: EMPEROR: A Multicenter, Randomized, Double-blind, Sham-controlled, Parallel Group, Phase 3 Study Evaluating the Efficacy, Safety, and Tolerability of Zorevunersen (STK-001) in Patients With Dravet Syndrome
Brief Title: A Double-blind Study Evaluating the Efficacy, Safety, and Tolerability of Zorevunersen in Patients With Dravet Syndrome
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Stoke Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STK-001-DS-301; 2024-519555-28 (EudraCT Number)
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Dravet Syndrome
Keywords: Pediatric epilepsy; Epileptic Encephalopathies; Refractory Myoclonic Epilepsy; Severe Myoclonic Epilepsy in Infancy; STK-001
MeSH Terms: conditions — Epilepsies, Myoclonic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zorevunersen (Experimental): Eligible patients will be randomly assigned in a 1:1 ratio to zorevunersen:sham in Treatment Period 1 (approximately 52 weeks). Upon the completion of Treatment Period 1 all eligible patients, will enter Treatment Period 2 and receive zorevunersen, regardless of initial treatment assignment.
  Interventions: Drug: zorevunersen
- Sham Comparator (Sham Comparator): Eligible patients will be randomly assigned in a 1:1 ratio to zorevunersen:sham
  Interventions: Other: Sham Comparator

INTERVENTIONS:
Drug: zorevunersen — Treatment Period 1: Zorevunersen group will receive study drug by intrathecal (IT) administration on Day 1 (after the 8-week Baseline Period), Day 57 (Week 8), Day 169 (Week 24), and Day 281 (Week 40) at a dose level of 70 mg on Day 1 and Day 57, and 45 mg on Day 169 and Day 281.
  Treatment Period 2: Group assigned to zorevunersen in Treatment Period 1 will receive 45 mg of zorevunersen on Day 393 (Week 56), Day 477 (Week 68), and Day 589 (Week 84).
  Arms: Zorevunersen
Other: Sham Comparator — Treatment Period 1: Sham group will not have drug administered. Sham group will have a procedure intended to mimic the drug administration.
  Treatment Period 2: Group assigned to sham in Treatment Period 1 will receive 70 mg of zorevunersen on Day 393 (Week 56) and on Day 477 (Week 68), and 45 mg of zorevunersen Day 589 (Week 84).
  Arms: Sham Comparator

SUMMARY:
The purpose of the study is to evaluate the efficacy, safety, and tolerability of zorevunersen in Patients with Dravet syndrome.

DETAILED DESCRIPTION:
Zorevunersen is an investigational new medicine for the treatment of Dravet syndrome. It is an antisense oligonucleotide (ASO) that is intended to increase the level of productive SCN1A messenger RNA (mRNA) and consequently increase the expression of the sodium channel Nav1.1 protein. This RNA-based approach is not gene therapy, but rather RNA modulation, as it does not manipulate nor insert genetic deoxyribonucleic acid (DNA).

Zorevunersen is designed to upregulate Nav1.1 protein expression from the nonmutant (wild-type) copy of the SCN1A gene to restore physiological Nav1.1 levels. Nav1.1 levels are reduced in people with Dravet syndrome.

This is a global, multicenter, randomized, double-blind, sham-controlled, parallel group Phase 3 study to assess the efficacy, safety, and tolerability of zorevunersen in patients with Dravet syndrome. The study duration and endpoints are designed to evaluate the potential of zorevunersen for disease modification. The study consists of two parts, Treatment Period 1 and Treatment Period 2. The primary and secondary endpoints will be assessed at the conclusion of Treatment Period 1. These endpoints will be assessed again at the end of Treatment Period 2. The primary endpoint is the change from baseline in major motor seizure frequency. Secondary endpoints include the change in behavior and cognition, clinical status, and health-related quality of life in patients with Dravet syndrome.

Patients will have the opportunity to enroll in an open label extension study and receive zorevunersen if they meet eligibility criteria at the end of the study.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patients must be ≥2 and <18 years of age.
2. Patients must have a clinical diagnosis of DS confirmed by the Epilepsy Study Consortium, Inc. (ESCI) and as defined by:

   Onset, prior to 12 months (inclusive, <13 months), of age, of recurrent focal with motor signs, hemiclonic, or generalized tonic-clonic seizures. No other known etiology causing clinical DS manifestations..
3. Patient must have a documented pathogenic, likely pathogenic variant, or variant of uncertain significance in the sodium voltage-gated channel type 1 alpha subunit (SCN1A) gene. Patients who have SCN1A testing results of Negative (no variants identified) cannot be randomized.
4. Patient must experience the required number of major motor seizures during the 6-week Observation Period. Major motor seizure types included are Seizure types included in counts are Hemiclonic, Focal with Motor Signs, Focal to Bilateral Tonic-Clonic, Generalized Tonic-Clonic, Tonic, Tonic/Atonic (Drop Attacks with fall or risk of fall), and Bilateral Clonic.
5. Patient must have used at least 2 prior interventions for seizures. These can include anti-seizure medications (ASMs), ketogenic diet and/or vagus nerve stimulation (VNS) with either lack of adequate seizure control or discontinued due to an AE(s). These interventions can be ongoing therapies.
6. Patient must be taking at least one ASM. Benzodiazepines or ASMs used on a standing basis (i.e., not as needed [PRN]) for any indication will be considered an ASM.
7. Patients' maintenance ASMs and interventions for seizures (i.e., ketogenic diet or VNS), as well as any marijuana- or cannabinoid-based products, must have been stable (unless adjusted for weight) during the Baseline Period.

Key Exclusion Criteria:

1. Patient has documented variant in the SCN1A gene associated with gain-of-function
2. Patient is currently treated with a maintenance ASM acting primarily as a sodium channel blocker, including but not limited to phenytoin, carbamazepine, oxcarbazepine, lamotrigine, lacosamide, rufinamide, or cenobamate, given the mechanism of action of zorevunersen.
3. Patient is currently treated with neuromodulation techniques (e.g., responsive neurostimulation, deep brain stimulation, or transcranial magnetic stimulation), with the exception of VNS.
4. Patient has emergence of a new seizure type or reemergence of a past seizure type (seizure types that last occurred more than 12 months before Screening Visit A) during the Baseline Period, or has more than 1 hospitalization for seizures during the Baseline Period.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 170 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Measurement of Seizure Change | Week 28
  Measured by daily seizure diary

SECONDARY OUTCOMES:
Measurement of Seizure Change | Week 52
  Measured by daily seizure diary
Multi-component Vineland Adaptive Behavior Scales, Third Edition (Vineland-3) Outcome Score | Week 52
  Measurement of change from baseline for multi-component score. Scoring is non-parametric and based on rank between treatment and sham groups. Individual items are scored on a scale of 0, 1, or 2, indicating never, sometimes, or usually or often, or on a scale of 0 or 2, indicating no or yes, with higher scores indicating greater performance
Vineland Adaptive Behavior Scales, Third Edition (Vineland-3) Subdomain Score | Week 52
  Measurement of change from baseline for individual subdomains. Scoring is point-based on a scale that varies, depending on subdomain, Individual items are scored on a scale of 0, 1, or 2, indicating never, sometimes, or usually or often, or on a scale of 0 or 2, indicating no or yes, with higher scores indicating greater performance.

CONTACTS AND LOCATIONS:
Locations (46):
- United States (32):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Cedars Sinai Medical Center, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - USCF Medical Center, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nemours Children's Health, Jacksonville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Advent Health Neuroscience Research Institute, Orlando, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - CS Mott Children's Hospital, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University in St. Louis School of Medicine, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - Weill Cornell Medicine, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Health System, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - LeBonheur Children's Hospital, Memphis, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Utah Primary Children's Hospital, Salt Lake City, Utah
  - UVA Health, Charlottesville, Virginia
- Japan (11):
  - Fukuoka Children's Hospital, Fukuoka
  - Hokkaido University Hospital, Hokkaido
  - Kyoto University Hospital, Kyoto
  - Nagoya University Hospital, Nagoya
  - National Hospital Organization Nishi Niigata Central Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Osaka City General Hospital, Osaka
  - Jichi Medical University Hospital, Shimotsuke
  - NHO Shizuoka, Shizuoka
  - National Center of Neurology and Psychiatry, Tokyo
  - Yokohama City University Medical Center, Yokohama
- United Kingdom (3):
  - Royal Hospital for Children, Glasgow
  - Great Ormond Street Hospital for Children, London
  - Sheffield Children's Hospital, Sheffield